CLINICAL TRIAL: NCT02429102
Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of MT-8554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MT-8554-E01
Record Dates: First submitted 2015-04-16; First posted 2015-04-29 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Phase 1; Healthy subjects; Pharmacokinetics of MT-8554

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single ascending dose, MT-8554 or Placebo (Experimental)
  Interventions: Drug: MT-8554; Drug: Placebo
- Multiple ascending dose, MT-8554 or Placebo (Experimental)
  Interventions: Drug: MT-8554; Drug: Placebo

INTERVENTIONS:
Drug: MT-8554
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of MT-8554 in healthy Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease
* Male or female subjects aged 18 to 55 years or elderly male subjects aged ≥65
* A body weight of ≥60 kg male and ≥50 kg female

Exclusion Criteria:

* Participation in more than three clinical studies involving administration of an Investigational Medicinal Product (IMP) in the previous year, or any study within 12 weeks.
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro-intestinal, renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness disorder.
* Clinically relevant abnormal medical history, physical findings or laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by vital signs | up to Day14
Safety and Tolerability as measured by ECG | up to Day14
Safety and Tolerability as measured by continuous lead II ECG monitoring | up to Day14
Safety and Tolerability as measured by laboratory safety assessments | up to Day14
Safety and Tolerability as measured by physical examination | up to Day14
Safety and Tolerability as measured by number of participants with adverse events | up to Day14

SECONDARY OUTCOMES:
PK profile (Cmax, tmax, t½, AUC) | 240 hours post dose
  Cmax, tmax, t½, AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational center, City Name, United Kingdom